CLINICAL TRIAL: NCT05536804
Title: Tirzepatide Study of Renal Function in People With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes: Focus on Kidney Hypoxia in Relation to Fatty Kidney Disease Using Multiparametric Magnetic Resonance Imaging
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes
Acronym: TREASURE-CKD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17217; I8F-MC-GPIG (Other: Eli Lilly and Company); 2021-005273-47 (EudraCT Number); 2023-506082-60-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Overweight; Obesity; Chronic Kidney Disease; Type 2 Diabetes; T2D
MeSH Terms: conditions — Overweight; Obesity; Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tirzepatide (Experimental): Tirzepatide administered subcutaneously (SC)
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Arms: Tirzepatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
We are doing this study to learn more about how tirzepatide may help fight chronic kidney disease in people with obesity with or without type 2 diabetes (T2D).

The study will last about 56 weeks and include up to 12 visits.

ELIGIBILITY:
Inclusion Criteria:

All participants with or without diabetes:

* Have a Body Mass Index (BMI) ≥27 kilogram/square meter (kg/m²) at screening
* Diagnosed with chronic kidney disease (CKD)
* Has an estimated glomerular filtration rate (eGFR) ≥25 to ≤60 ml/min/1.73 m² or eGFR ≥25 to ≤75 ml/min/1.73 m² if urine albumin-to-creatinine ratio (UACR) >30 milligram/gram (mg/g)
* Have been receiving an angiotensin-converting enzyme (ACE) or angiotensin II receptor blockers (ARB) that is considered the maximal appropriate dose by the investigator for treatment of chronic kidney disease or hypertension (unless the participant has low blood pressure or hypotension)

Participants without diabetes:

* Have Hemoglobin A1c (HbA1c) <6.5% at screening

Participants with Type 2 diabetes:

* Have been diagnosed at least 180 days prior to screening
* Have HbA1c ≤9.5% at screening

Exclusion Criteria:

All participants:

* Have a self-reported change in body weight >5 kilogram (kg) within 90 days prior to screening.
* Have a prior or planned surgical treatment for obesity
* Have or plan to have endoscopic and/or device-based therapy for obesity or have had device removal within the last 180 days
* Have eGFR <25 mL/min/1.73m² calculated by using creatinine-based chronic kidney disease epidemiology collaboration (CKD-EPI) equations, as determined by central laboratory at screening.
* Have a history of unstable or rapidly progressing renal disease according to investigator judgment
* Have a known clinically significant gastric emptying abnormality (for example, severe diabetic gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect GI motility)
* Have had a history of chronic or acute pancreatitis

Participants with T2D:

* Have history of proliferative diabetic retinopathy or diabetic macular edema or non-proliferative diabetic retinopathy that requires acute treatment.
* Have been diagnosed with type 1 diabetes (T1D) or have history of ketoacidosis or hyperosmolar state/coma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Kidney Oxygenation in Participants With or Without T2D | Baseline, Week 52
  Blood oxygenation-level dependent magnetic resonance imaging (BOLD MRI)

SECONDARY OUTCOMES:
Change from Baseline in Kidney Oxygenation in Participants with T2D (BOLD MRI) | Baseline, Week 52
Change from Baseline in Kidney Oxygenation in Participants without T2D (BOLD MRI) | Baseline, Week 52
Percent Change from Baseline in Body Weight | Baseline, Week 52
Percent Change from Baseline in Renal Sinus Fat Content (MRI) | Baseline, Week 52
Percent Change from Baseline in Renal Fat Content (MRI Proton Density Fat Fraction) | Baseline, Week 52
Percent Change from Baseline in Renal Blood Flow (Phase-Contrast MRI) | Baseline, Week 52
Change from Baseline in Apparent Diffusion Coefficient (ADC) MRI | Baseline, Week 52
Change from Baseline in Glomerular Filtration Rate (GFR) Iohexol Clearance in Milliliter/Minute/Square Meter (ml/min/m²) | Baseline, Week 52
Change from Baseline in 24-hour Urinary Albumin Excretion (UAE) in Milligram/24 Hours (mg/24h) | Baseline, Week 52
Percent Change from Baseline in Urine Albumin-to-Creatine Ratio (UACR) | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (27):
- United States (10):
  - Valley Clinical Trials, Inc., Northridge, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Kidney Associates of Colorado, Denver, Colorado
  - American Health Network of Indiana, LLC - Avon, Avon, Indiana
  - American Health Network of Indiana, LLC - Greenfield, Greenfield, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - American Health Network of Indiana, LLC - Muncie, Muncie, Indiana
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Providence Medical Research Center - Spokane, Spokane, Washington
- Austria (3):
  - Klinik Landstraße, Vienna
  - Zentrum für klinische Studien Dr Hanusch Gmbh, Vienna
  - Klinik Hietzing, Vienna
- Canada (5):
  - LMC Clinical Research Inc. (Barrie), Barrie
  - LMC Clinical Research Inc. (Thornhill), Concord
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie Centre Hospitalier Universitaire -T, Sherbrooke
  - Toronto General Hospital, Toronto
  - Fadia El Boreky Medicine, Waterloo
- Aarhus Universitetshospital, Skejby, Aarhus, Denmark
- Mexico (6):
  - Centro de Investigación y Gastroenterología, Cuauhtémoc
  - Investigación Nefrológica, Cuernavaca
  - Health Pharma Professional Research S.A. de C.V:, Mexico City
  - Grupo Medico Camino Sc, Mexico City
  - Caimed Investigacion En Salud S.A. de C.V., Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, México
- Netherlands (2):
  - Ziekenhuisgroep Twente, locatie Almelo, Almelo
  - Amsterdam UMC, locatie VUmc, Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Heerspink HJL, Friedman AN, Bjornstad P, van Raalte DH, Cherney D, Cao D, Garcia-Perez LE, Stefanski A, Turfanda I, Bunck MC, Benabbad I, Griffin R, Piras de Oliveira C. Kidney Parameters with Tirzepatide in Obesity with or without Type 2 Diabetes. J Am Soc Nephrol. 2025 Nov 1;36(11):2190-2200. doi: 10.1681/ASN.0000000764. Epub 2025 Jun 13. PMID 40512543
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: A Study of Tirzepatide (LY3298176) in Participants With Overweight or Obesity and Chronic Kidney Disease With or Without Type 2 Diabetes (TREASURE-CKD) — https://trials.lilly.com/en-US/trial/360461